CLINICAL TRIAL: NCT01089400
Title: Immuno-virological Characterization of Severe H1N1v Influenza Infection in Bronchoalveolar Lavage in Patients Requiring Mechanical Ventilation in Intensive Care Unit
Brief Title: Immuno-virological Characterization of Severe H1N1v Influenza Infection in Bronchoalveolar Lavage
Acronym: FluBAL
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: C09-39
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2012-01

CONDITIONS: Influenza; Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: influenza; H1N1; lymphocytes; T cell; CD4; CD8; cytokine; serology; broncho-alveolar lavage; acute respiratory distress syndrome; ventilation; intensive care unit
MeSH Terms: conditions — Influenza, Human; Acute Lung Injury; Respiratory Distress Syndrome; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchoalveolar lavage fuid Nasal sample Peripheral mononuclear blood cells Plasma Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Influenza A/H1N1 patients
- Non influenza A/H1N1 patients

SUMMARY:
The influenza A/H1N1v pandemic virus causes severe pneumonia that can lead to acute respiratory distress syndrome and death even in healthy young individuals. The respective roles of viral replication, bacterial infection and immune alterations of the host during such severe influenza H1N1v infection need to be clarified in order to optimize patients care. In this context, we aim to study immune and virological parameters in bronchoalveolar lavage fluid during severe influenza A/H1N1v infection with pulmonary involvement in intensive care unit. Results will be correlated to bacterial or viral pulmonary co-infections and to peripheral blood immune and virological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Suspected influenza A/H1N1 infection
* Diffuse bilateral pneumonia <96h with acute lung injury or respiratory distress syndrome
* Invasive or non-invasive ventilation in intensive care unit
* Age > 13

Exclusion Criteria:

* Other cause identified of acute lung injury or acute respiratory distress syndrome
* Contraindicated bronchoalveolar lavage

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe influenza A/H1N1v infection with pulmonary involvement in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
immunological parameters in blood and bronchoalveolar lavage fluid | day 0 and day 5-7 of ventilation for both blood and BAL, day 30 and month 5 for blood

SECONDARY OUTCOMES:
virological parameters in nose, broncho-alveolar lavage and peripheral blood | day 0 and day 5-7 of ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Guihot, MD PhD, Principal Investigator — INSERM UMR945
Locations (2):
- France (2):
  - Pitie-Salpetrière Hospital, Paris
  - Tenon Hospital, Paris

REFERENCES:
- [Result] Guihot A, Luyt CE, Parrot A, Rousset D, Cavaillon JM, Boutolleau D, Fitting C, Pajanirassa P, Mallet A, Fartoukh M, Agut H, Musset L, Zoorob R, Kirilovksy A, Combadiere B, van der Werf S, Autran B, Carcelain G; FluBAL Study Group. Low titers of serum antibodies inhibiting hemagglutination predict fatal fulminant influenza A(H1N1) 2009 infection. Am J Respir Crit Care Med. 2014 May 15;189(10):1240-9. doi: 10.1164/rccm.201311-2071OC. PMID 24646009